CLINICAL TRIAL: NCT00381797
Title: Phase II Study of Bevacizumab Plus Irinotecan (Camptosar™) in Children With Recurrent, Progressive, or Refractory Malignant Gliomas, Diffuse/Intrinsic Brain Stem Gliomas, Medulloblastomas, Ependymomas and Low Grade Gliomas
Brief Title: Bevacizumab and Irinotecan in Treating Young Patients With Recurrent, Progressive, or Refractory Glioma, Medulloblastoma, Ependymoma, or Low Grade Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-01090; NCI-2009-01090 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PBTC-022; CDR0000499832; PBTC-022 (Other: Pediatric Brain Tumor Consortium); PBTC-022 (Other: CTEP); U01CA081457 (NIH)
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Results first posted 2013-01-15 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-10

CONDITIONS: Childhood Cerebral Anaplastic Astrocytoma; Childhood Oligodendroglioma; Childhood Spinal Cord Neoplasm; Recurrent Childhood Brain Stem Glioma; Recurrent Childhood Ependymoma; Recurrent Childhood Medulloblastoma
MeSH Terms: conditions — Oligodendroglioma; Spinal Cord Neoplasms; Familial ependymoma; Medulloblastoma | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Fluorodeoxyglucose F18; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15 and irinotecan hydrochloride IV over 90 minutes on day 16 or 17 for course 1. Patients receive bevacizumab and irinotecan hydrochloride on days 1 and 15 for all subsequent courses. Treatment repeats every 4 weeks for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Patients undergo MRIs of the brain, magnetic resonance perfusion/diffusion, and fludeoxyglucose F 18 positron emission tomography at baseline and periodically during treatment.
  Interventions: Biological: Bevacizumab; Radiation: Fludeoxyglucose F-18; Drug: Irinotecan Hydrochloride

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar FKB238; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
Radiation: Fludeoxyglucose F-18 — Undergo fludeoxyglucose F18 PET
  Other Names: 18FDG; FDG; fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; Irinomedac; U-101440E

SUMMARY:
This phase II trial is studying how well giving bevacizumab together with irinotecan works in treating young patients with recurrent, progressive, or refractory glioma, medulloblastoma, ependymoma, or low grade glioma. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of glioma by blocking blood flow to the tumor. Drugs used in chemotherapy, such as irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bevacizumab together with irinotecan may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Estimate the rates of objective response observed prior to disease progression during the first four courses of treatment with bevacizumab and irinotecan hydrochloride in pediatric patients with recurrent, progressive, or refractory malignant glioma (Stratum A [closed to accrual as of 4/21/2009]) or recurrent/progressive/refractory intrinsic brain stem glioma (Stratum B [closed to accrual as of 4/21/2009]).

II. Estimate the rates of objective response observed prior to disease progression during the first four courses of treatment with bevacizumab and irinotecan hydrochloride in patients with recurrent or progressive medulloblastoma (Stratum C [closed to accrual as of 10/27/2009]) or recurrent or progressive ependymoma (Stratum D [closed to accrual as of 7/29/2010]).

III. Estimate the sustained disease stabilization rate associated with bevacizumab and irinotecan in patients with recurrent or progressive low grade glioma (Stratum E [closed to accrual as of 7/29/2010]).

SECONDARY OBJECTIVES:

I. Estimate the rate of treatment-related toxicity of this regimen in these patients.

II. Estimate the cumulative incidence of sustained objective responses as a function of this regimen in these patients.

III. Estimate the distributions of survival and event-free survival of these patients.

IV. Correlate functional changes in tumor with progression-free survival and response using MR perfusion/diffusion imaging and fludeoxyglucose F 18 positron emission tomography.

OUTLINE: This is a multicenter study. Patients are stratified according to tumor type (high-grade glioma [closed to accrual as of 4/21/2009] vs intrinsic brain stem tumor [closed to accrual as of 4/21/2009] vs medulloblastoma [closed to accrual as of 10/27/2010] vs ependymoma [closed to accrual as of 7/29/2010] vs low grade glioma [closed to accrual as of 7/29/2010]).

Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15 and irinotecan hydrochloride IV over 90 minutes on day 16 or 17 for course 1. Patients receive bevacizumab and irinotecan hydrochloride on days 1 and 15 for all subsequent courses. Treatment repeats every 4 weeks for up to 24 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo MRIs of the brain, magnetic resonance perfusion/diffusion, and fludeoxyglucose F 18 positron emission tomography at baseline and periodically during treatment.

After completion of study treatment, patients are followed for 30 days and then every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed high-grade glioma (WHO grade III or IV) at any site within the brain, including the following:

  * Anaplastic astrocytoma
  * Glioblastoma multiforme (including giant cell and gliosarcoma subtypes)
  * Anaplastic oligodendroglioma
  * Anaplastic ganglioglioma
  * Anaplastic oligoastrocytoma
  * Diffuse brain stem glioma

    * Histologic confirmation not required
  * Histologically confirmed medulloblastoma
  * Histologically confirmed ependymoma
  * Primary spinal cord malignant glioma with measurable metastatic disease within the brain

    * Histologic confirmation required
    * Neuraxis dissemination allowed provided there is bidimensionally measurable disease within the brain and spinal cord
  * Low grade glioma at any site within the brain with or without spinal cord disease
* Recurrent, progressive, or refractory disease (must have received prior chemoradiotherapy)
* No more than 2 prior chemotherapy regimens following relapse
* Bidimensionally measurable disease, defined as ≥ 1 lesion that can be accurately measured in ≥ 2 planes
* If there is spinal cord disease as well, response assessment will be based only upon the measurable tumor in the brain
* No diffuse gliomatosis cerebri with < 1 discrete, measurable lesion
* No evidence of new symptomatic CNS hemorrhage (> grade 2) within the past 2 weeks
* No central non-cerebellar PNET's (e.g., cerebral PNET or pineoblastoma)
* No spinal cord tumors only
* Karnofsky performance status (PS) 50-100% (> 16 years of age) OR Lansky PS 50-100% (≤ 16 years of age)
* Absolute neutrophil count ≥ 1,500/mm³ (unsupported)
* Platelet count ≥ 100,000/mm³ (unsupported)
* Hemoglobin > 8 g/dL (support allowed)
* Creatinine normal
* BUN < 25 mg/dL
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT and AST ≤ 3 times ULN
* Neurological deficits must be stable for ≥ 1 week prior to study entry
* No active renal, cardiac (congestive cardiac failure, myocarditis), or pulmonary disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 6 months after completion of study treatment
* No clinically significant unrelated systemic illness that would preclude study treatment, including any of the following:

  * Serious infections
  * Significant cardiac, pulmonary, hepatic, or other organ dysfunction
  * No uncontrolled systemic hypertension, defined as systolic blood pressure (BP) and/or diastolic BP > 95th percentile for age
  * No stroke, myocardial infarction, or unstable angina within the past 6 months
  * No clinically significant peripheral vascular disease
  * No significant traumatic injury within the past 6 weeks
  * No evidence of bleeding diathesis, coagulopathy, or PT INR > 1.5
  * Urine protein/creatinine ratio ≤ 1.0
  * No abdominal fistula or gastrointestinal perforation within the past 6 months
  * No serious nonhealing wound, ulcer, or bone fracture
* At least 3 weeks since prior myelosuppressive anticancer chemotherapy (6 weeks for nitrosoureas)
* At least 7 days since prior investigational or biologic agents (3 weeks if patient experienced ≥ grade 2 myelosuppression or if agent has a prolonged half-life)
* More than 7 days since prior minor surgery
* More than 12 weeks since prior craniospinal or focal irradiation to primary tumor or other sites
* At least 4 weeks since prior major surgery and recovered
* At least 3 months since prior autologous bone marrow or stem cell transplantation
* At least 2 weeks since prior colony-forming growth factors (i.e., filgrastim [G-CSF], sargramostim [GM-CSF], epoetin alfa)
* No prior bevacizumab or irinotecan hydrochloride
* No anticipated surgery during treatment
* No concurrent prophylactic G-CSF, GM-CSF, or epoetin alfa
* Concurrent dexamethasone allowed provided the dose is stable or decreasing over the past week
* No other concurrent anticancer or investigational drugs
* No concurrent medications that may interfere with study (e.g., immunosuppressive agents other than corticosteroids)
* No concurrent therapeutic anticoagulation
* No concurrent nonsteroidal anti-inflammatory drugs, clopidogrel bisulfate, dipyridamole, or acetylsalicylic acid (aspirin) > 81 mg/day

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 97 (Actual)
Dates: Start 2006-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sridharan Gururangan, Principal Investigator — Pediatric Brain Tumor Consortium
Locations (11):
- United States (11):
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Pediatric Brain Tumor Consortium, Memphis, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Background] Han K, Peyret T, Quartino A, Gosselin NH, Gururangan S, Casanova M, Merks JH, Massimino M, Grill J, Daw NC, Navid F, Jin J, Allison DE. Bevacizumab dosing strategy in paediatric cancer patients based on population pharmacokinetic analysis with external validation. Br J Clin Pharmacol. 2016 Jan;81(1):148-60. doi: 10.1111/bcp.12778. Epub 2015 Dec 10. PMID 26345283
- See also: Bevacizumab dosing strategy in paediatric cancer patients based on population pharmacokinetic analysis with external validation — https://www.ncbi.nlm.nih.gov/pubmed/26345283

RESULTS

PARTICIPANT FLOW:
Groups:
- High-grade Gliomas: Recurrent, progressive or refractory high-grade gliomas (Stratum A): The only patients with Recurrent, progressive or refractory high-grade gliomas were treated in this arm. Therapy will begin with single-agent bevacizumab 10 mg/kg given intravenously (i.v) on day 1 and day 15 (+/- 24 hours) followed by MR-perfusion/diffusion imaging within 24-48 hours following the 2nd dose of bevacizumab. The first dose of irinotecan will be given i.v following this MR-perfusion scan. Subsequently, bevacizumab and irinotecan will be given every two weeks. The irinotecan dose will depend on whether the patient is on an enzyme-inducing anticonvulsant drug (EIACD). The irinotecan dose will be 250 mg/m2 (~ 80 % of dose tolerated by adults in the Duke Phase II study of bevacizumab plus irinotecan) every two weeks for those on EIACDs. If the patient is not on an EIACD, the starting dose will be 125 mg/m2.
- Brain Stem Tumors: Recurrent,progressive or refractory intrinsic brain stem tumors (Stratum B): The only patients with Recurrent,progressive or refractory intrinsic brain stem tumors were treated in this arm. Therapy will begin with single-agent bevacizumab 10 mg/kg given intravenously (i.v) on day 1 and day 15 (+/- 24 hours) followed by MR-perfusion/diffusion imaging within 24-48 hours following the 2nd dose of bevacizumab. The first dose of irinotecan will be given i.v following this MR-perfusion scan. Subsequently, bevacizumab and irinotecan will be given every two weeks. The irinotecan dose will depend on whether the patient is on an enzyme-inducing anticonvulsant drug (EIACD). The irinotecan dose will be 250 mg/m2 (~ 80 % of dose tolerated by adults in the Duke Phase II study of bevacizumab plus irinotecan) every two weeks for those on EIACDs. If the patient is not on an EIACD, the starting dose will be 125 mg/m2.
- Medulloblastoma: Recurrent or progressive medulloblastoma(Stratum C): The only patients with recurrent or progressive medulloblastoma were treated in this arm. Therapy will begin with single-agent bevacizumab 10 mg/kg given intravenously (i.v) on day 1 and day 15 (+/- 24 hours) followed by MR-perfusion/diffusion imaging within 24-48 hours following the 2nd dose of bevacizumab. The first dose of irinotecan will be given i.v following this MR-perfusion scan. Subsequently, bevacizumab and irinotecan will be given every two weeks. The irinotecan dose will depend on whether the patient is on an enzyme-inducing anticonvulsant drug (EIACD). The irinotecan dose will be 250 mg/m2 (~ 80 % of dose tolerated by adults in the Duke Phase II study of bevacizumab plus irinotecan) every two weeks for those on EIACDs. If the patient is not on an EIACD, the starting dose will be 125 mg/m2.
- Ependymoma: Recurrent or progressive ependymoma (Stratum D):The only patients with recurrent or progressive ependymoma were treated in this arm. Therapy will begin with single-agent bevacizumab 10 mg/kg given intravenously (i.v) on day 1 and day 15 (+/- 24 hours) followed by MR-perfusion/diffusion imaging within 24-48 hours following the 2nd dose of bevacizumab. The first dose of irinotecan will be given i.v following this MR-perfusion scan. Subsequently, bevacizumab and irinotecan will be given every two weeks. The irinotecan dose will depend on whether the patient is on an enzyme-inducing anticonvulsant drug (EIACD). The irinotecan dose will be 250 mg/m2 (~ 80 % of dose tolerated by adults in the Duke Phase II study of bevacizumab plus irinotecan) every two weeks for those on EIACDs. If the patient is not on an EIACD, the starting dose will be 125 mg/m2.
- Low Grade Glioma: Recurrent low grade glioma (Stratum E): The only patients with recurrent low grade glioma were treated in this arm. Therapy will begin with single-agent bevacizumab 10 mg/kg given intravenously (i.v) on day 1 and day 15 (+/- 24 hours) followed by MR-perfusion/diffusion imaging within 24-48 hours following the 2nd dose of bevacizumab. The first dose of irinotecan will be given i.v following this MR-perfusion scan. Subsequently, bevacizumab and irinotecan will be given every two weeks. The irinotecan dose will depend on whether the patient is on an enzyme-inducing anticonvulsant drug (EIACD). The irinotecan dose will be 250 mg/m2 (~ 80 % of dose tolerated by adults in the Duke Phase II study of bevacizumab plus irinotecan) every two weeks for those on EIACDs. If the patient is not on an EIACD, the starting dose will be 125 mg/m2.
Period: Overall Study
Arm/Group | High-grade Gliomas | Brain Stem Tumors | Medulloblastoma | Ependymoma | Low Grade Glioma
Started | 18 | 17 | 10 | 15 | 37
Completed | 17 | 16 | 10 | 14 | 35
Not Completed | 1 | 1 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 2
Not completed — Ineligible | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High-grade Gliomas | Brain Stem Tumors | Medulloblastoma | Ependymoma | Low Grade Glioma | Total
Number analyzed (Participants) | 18 | 17 | 10 | 15 | 37 | 97
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 17 | 9 | 14 | 37 | 91
  Between 18 and 65 years | 4 | 0 | 1 | 1 | 0 | 6
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.07 (3.82) | 8.45 (3.35) | 10.56 (5.28) | 10.16 (5.17) | 8.58 (4.09) | 10.21 (4.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 5 | 9 | 19 | 49
  Male | 11 | 8 | 5 | 6 | 18 | 48
Region of Enrollment [Number; unit: participants]
  United States | 18 | 17 | 10 | 15 | 37 | 97

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate Sustained for ≥ 8 Weeks
Description: Objective response is either a complete response or a partial response observed during the first four courses of treatment and sustained for 8 weeks. The objective response rate will be reported separately for patients with recurrent/progressive malignant glioma(Stratum A), recurrent/progressive instrinsic brain stem tumors(Stratum B), recurrent/progressive medulloblastoma(Stratum C), and recurrent/progressive ependymoma(Stratum D). CR is complete disappearance of all enhancing tumor. PR is >= 50% reduction in tumor size. This outcome measures is not defined for the Stratum E in the protocol.
Time Frame: From day 1 of treatment up to 24 weeks
Population: Two patients in the Stratum A,one patient in the Stratum C, and one patient in the Stratum D were inevaluable for this outcome measure.
Measure: Number; unit: participants
Groups:
- Brain Stem Tumors: Recurrent, progressive or refractory intrinsic brain stem tumors (Stratum B):The only patients with recurrent, progressive or refractory brain stem tumors were treated in this arm. Therapy will begin with single-agent bevacizumab 10 mg/kg given intravenously (i.v) on day 1 and day 15 (+/- 24 hours) followed by MR-perfusion/diffusion imaging within 24-48 hours following the 2nd dose of bevacizumab. The first dose of irinotecan will be given i.v following this MR-perfusion scan. Subsequently, bevacizumab and irinotecan will be given every two weeks. The irinotecan dose will depend on whether the patient is on an enzyme-inducing anticonvulsant drug (EIACD). The irinotecan dose will be 250 mg/m2 (~ 80 % of dose tolerated by adults in the Duke Phase II study of bevacizumab plus irinotecan) every two weeks for those on EIACDs. If the patient is not on an EIACD, the starting dose will be 125 mg/m2.
- Medulloblastoma: Recurrent or progressive medulloblastoma(Stratum C):The only patients with recurrent or progressive medulloblastoma were treated in this arm. Therapy will begin with single-agent bevacizumab 10 mg/kg given intravenously (i.v) on day 1 and day 15 (+/- 24 hours) followed by MR-perfusion/diffusion imaging within 24-48 hours following the 2nd dose of bevacizumab. The first dose of irinotecan will be given i.v following this MR-perfusion scan. Subsequently, bevacizumab and irinotecan will be given every two weeks. The irinotecan dose will depend on whether the patient is on an enzyme-inducing anticonvulsant drug (EIACD). The irinotecan dose will be 250 mg/m2 (~ 80 % of dose tolerated by adults in the Duke Phase II study of bevacizumab plus irinotecan) every two weeks for those on EIACDs. If the patient is not on an EIACD, the starting dose will be 125 mg/m2.
Arm/Group | High-grade Gliomas | Brain Stem Tumors | Medulloblastoma | Ependymoma
Number analyzed (Participants) | 15 | 16 | 9 | 13
participants | 0 | 0 | 0 | 0

2. Primary Outcome: Sustained Disease Stabilization Rate Associated With Bevacizumab and Irinotecan in Patients With Recurrent or Progressive Low-grade Glioma (Stratum E)
Description: Disease stabilization is defined as a complete response(CR) or partial response(PR) observed during the first four courses and sustained for 8 weeks; or stable disease (SD) sustained for 6 courses characterized by SD at the end of course 2, at the end of course 4 and at the end of course 6. CR is complete disappearance of all enhancing tumor. PR is >= 50% reduction in tumor size. SD is at least stable and maintenance corticosteroid dose not increased in neurologic examination.
Time Frame: From day 1 of treatment up to 24 weeks
Population: Patients with recurrent or progressive low grade glioma were treated with any courses.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Low Grade Glioma
Number analyzed (Participants) | 35
participants | 23 [17 to 28]

3. Secondary Outcome: Number of Study Participants With Grade 3 or 4 Treatment-related Toxicity
Description: Adverse events are monitored and graded according to the Common Terminology Criteria for Adverse Events. The grade 1 = mild, grade 2=moderate, grade 3 =severe, grade 4=life threatening/disabling, grade 5=death.
Time Frame: From day 1 of treatment until off study
Population: The patients were treated with any dose treatment.
Measure: Number; unit: participants
Groups:
- High-grade Gliomas: Recurrent, progressive or refractory high-grade gliomas(Stratum A): The only patients with recurrent, progressive or refractory high-grade gliomas were treated in this arm. Therapy will begin with single-agent bevacizumab 10 mg/kg given intravenously (i.v) on day 1 and day 15 (+/- 24 hours) followed by MR-perfusion/diffusion imaging within 24-48 hours following the 2nd dose of bevacizumab. The first dose of irinotecan will be given i.v following this MR-perfusion scan. Subsequently, bevacizumab and irinotecan will be given every two weeks. The irinotecan dose will depend on whether the patient is on an enzyme-inducing anticonvulsant drug (EIACD). The irinotecan dose will be 250 mg/m2 (~ 80 % of dose tolerated by adults in the Duke Phase II study of bevacizumab plus irinotecan) every two weeks for those on EIACDs. If the patient is not on an EIACD, the starting dose will be 125 mg/m2.
- Brain Stem Tumors: Recurrent, progressive or refractory intrinsic brain stem tumors(Stratum B):The only patients with recurrent, progressive or refractory brain stem tumors were treated in this arm. Therapy will begin with single-agent bevacizumab 10 mg/kg given intravenously (i.v) on day 1 and day 15 (+/- 24 hours) followed by MR-perfusion/diffusion imaging within 24-48 hours following the 2nd dose of bevacizumab. The first dose of irinotecan will be given i.v following this MR-perfusion scan. Subsequently, bevacizumab and irinotecan will be given every two weeks. The irinotecan dose will depend on whether the patient is on an enzyme-inducing anticonvulsant drug (EIACD). The irinotecan dose will be 250 mg/m2 (~ 80 % of dose tolerated by adults in the Duke Phase II study of bevacizumab plus irinotecan) every two weeks for those on EIACDs. If the patient is not on an EIACD, the starting dose will be 125 mg/m2.
- Ependymoma: Recurrent or progressive ependymoma(Stratum D): The only patients with recurrent or progressive ependymoma were treated in this arm. Therapy will begin with single-agent bevacizumab 10 mg/kg given intravenously (i.v) on day 1 and day 15 (+/- 24 hours) followed by MR-perfusion/diffusion imaging within 24-48 hours following the 2nd dose of bevacizumab. The first dose of irinotecan will be given i.v following this MR-perfusion scan. Subsequently, bevacizumab and irinotecan will be given every two weeks. The irinotecan dose will depend on whether the patient is on an enzyme-inducing anticonvulsant drug (EIACD). The irinotecan dose will be 250 mg/m2 (~ 80 % of dose tolerated by adults in the Duke Phase II study of bevacizumab plus irinotecan) every two weeks for those on EIACDs. If the patient is not on an EIACD, the starting dose will be 125 mg/m2.
- Low Grade Glioma: Recurrent or progressive low grade glioma(Stratum E):The only patients with recurrent or progressive low grade glioma were treated in this arm. Therapy will begin with single-agent bevacizumab 10 mg/kg given intravenously (i.v) on day 1 and day 15 (+/- 24 hours) followed by MR-perfusion/diffusion imaging within 24-48 hours following the 2nd dose of bevacizumab. The first dose of irinotecan will be given i.v following this MR-perfusion scan. Subsequently, bevacizumab and irinotecan will be given every two weeks. The irinotecan dose will depend on whether the patient is on an enzyme-inducing anticonvulsant drug (EIACD). The irinotecan dose will be 250 mg/m2 (~ 80 % of dose tolerated by adults in the Duke Phase II study of bevacizumab plus irinotecan) every two weeks for those on EIACDs. If the patient is not on an EIACD, the starting dose will be 125 mg/m2.
Arm/Group | High-grade Gliomas | Brain Stem Tumors | Medulloblastoma | Ependymoma | Low Grade Glioma
Number analyzed (Participants) | 17 | 16 | 10 | 14 | 35
participants | 8 | 4 | 4 | 6 | 22

4. Secondary Outcome: Cumulative Incidence of Sustained Objective Responses
Description: Cumulative incidence of sustained objective response provides a percentage of participants experiencing the event of interest at a given follow-up time point (for example, 6-months, 1-year, etc.) in the presence of competing events such as progressive disease or death, and it is estimated using the event data for both the event of interest and the competing events experienced by the study participants. In this sense, it is different than the incidence rates estimated in epidemiological studies in terms of 'incidences per 1000 person years. 6-month Cumulative incidence of sustained objective responses will be reported separately for each stratum.
Time Frame: From the first imaging after treatment up to 2 years
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Groups:
- High-grade Gliomas: Recurrent, progressive or refractory high-grade gliomas(Stratum A):The only patients with Recurrent, progressive or refractory high-grade gliomas were treated in this arm. Therapy will begin with single-agent bevacizumab 10 mg/kg given intravenously (i.v) on day 1 and day 15 (+/- 24 hours) followed by MR-perfusion/diffusion imaging within 24-48 hours following the 2nd dose of bevacizumab. The first dose of irinotecan will be given i.v following this MR-perfusion scan. Subsequently, bevacizumab and irinotecan will be given every two weeks. The irinotecan dose will depend on whether the patient is on an enzyme-inducing anticonvulsant drug (EIACD). The irinotecan dose will be 250 mg/m2 (~ 80 % of dose tolerated by adults in the Duke Phase II study of bevacizumab plus irinotecan) every two weeks for those on EIACDs. If the patient is not on an EIACD, the starting dose will be 125 mg/m2.
- Low Grade Glioma: Recurrent or progressive low grade glioma(Stratum E): The only patients with Recurrent or progressive low grade glioma were treated in this arm. Therapy will begin with single-agent bevacizumab 10 mg/kg given intravenously (i.v) on day 1 and day 15 (+/- 24 hours) followed by MR-perfusion/diffusion imaging within 24-48 hours following the 2nd dose of bevacizumab. The first dose of irinotecan will be given i.v following this MR-perfusion scan. Subsequently, bevacizumab and irinotecan will be given every two weeks. The irinotecan dose will depend on whether the patient is on an enzyme-inducing anticonvulsant drug (EIACD). The irinotecan dose will be 250 mg/m2 (~ 80 % of dose tolerated by adults in the Duke Phase II study of bevacizumab plus irinotecan) every two weeks for those on EIACDs. If the patient is not on an EIACD, the starting dose will be 125 mg/m2.
Arm/Group | High-grade Gliomas | Brain Stem Tumors | Medulloblastoma | Ependymoma | Low Grade Glioma
Number analyzed (Participants) | 15 | 16 | 9 | 13 | 35
Percentage of Participants | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0.058 (0.0405)

5. Secondary Outcome: Progression-free Survival
Description: Progression-Free survival is the interval of time between of protocol treatment and minimum date of documentation of progressive Disease,second malignancy,death due to any cause, or date of last follow-up. Progressive neurologic abnormalities or worsening neurologic status not explained by causes unrelated to tumor progression,OR the appearance of new tumor OR a > 25% increase in the sum of the products of two longest perpendicular diameters of all measurable tumors. K-M method was used to estimate progression-free survival.
Time Frame: From start of treatment up to 2 years
Population: The patients were treated with any dose treatment.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Ependymoma: Recurrent or progressive ependymoma(Stratum D): The only patients with Recurrent, progressive ependymoma were treated in this arm. Therapy will begin with single-agent bevacizumab 10 mg/kg given intravenously (i.v) on day 1 and day 15 (+/- 24 hours) followed by MR-perfusion/diffusion imaging within 24-48 hours following the 2nd dose of bevacizumab. The first dose of irinotecan will be given i.v following this MR-perfusion scan. Subsequently, bevacizumab and irinotecan will be given every two weeks. The irinotecan dose will depend on whether the patient is on an enzyme-inducing anticonvulsant drug (EIACD). The irinotecan dose will be 250 mg/m2 (~ 80 % of dose tolerated by adults in the Duke Phase II study of bevacizumab plus irinotecan) every two weeks for those on EIACDs. If the patient is not on an EIACD, the starting dose will be 125 mg/m2.
Arm/Group | High-grade Gliomas | Brain Stem Tumors | Medulloblastoma | Ependymoma
Number analyzed (Participants) | 17 | 16 | 10 | 14
Months | 4.20 (1.57) [1.82 to 7.44] | 2.35 [1.85 to 4.17] | 2.48 [0.43 to 16.66] | 2.15 [1.85 to 6.15]

6. Secondary Outcome: Change in Perfusion Ratio Between the Baseline and Day 15 Brain Imaging
Description: Perfusion ratio obtained from magnetic resonance(MR) diffusion imaging may explain changes in the tumor after therapy. Changes in the perfusion ratio will be reported for those strata that have a sufficient number of participants with MR diffusion imaging. The change was calculated from perfusion ratio at Baseline to perfusion ratio at Day 15(values of perfusion ratio at Day 15 - values of perfusion ratio at baseline). The higher of perfusion ratio is worse.
  MR perfusion ratio is perfusion solid part of tumor from CBV divided by perfusion frontal while matter. There is no a unit available.
Time Frame: Baseline and day 15
Population: There are no sufficient data for the analyses in the Medulloblastoma arm and Ependymoma arm.
Measure: Median (Full Range); unit: Ratio
Arm/Group | High-grade Gliomas | Brain Stem Tumors | Low Grade Glioma
Number analyzed (Participants) | 9 | 5 | 19
Ratio | -0.14 (0.705) [-3.95 to 3.37] | -1.98 [-4.34 to -0.018] | -0.42 [-2.34 to 2.55]

7. Secondary Outcome: Change in Diffusion Ratio Between the Baseline and Day 15 Brain Image
Description: Diffusion ratio obtained from magnetic resonance (MR) diffusion imaging may explain changes in the tumor after therapy. Changes in the diffusion ratio will be reported for those strata that have a sufficient number of participants with MR diffusion imaging. The change was calculated from diffusion ratio at Baseline to diffusion ratio at Day 15 (values of diffusion ratio at Day 15 -values of diffusion ration at baseline). The higher of diffusion ratio is better. MR diffusion ratio is the diffusion solid part of tumor divided by the diffusion frontal white matter. There is no a unit available.
Time Frame: Baseline and day 15
Population: There are no sufficient data for the analyses in the Medulloblastoma arm.
Measure: Median (Full Range); unit: Ratio
Groups:
- Ependymoma: Recurrent or progressive ependymoma(Stratum D):The only patients with Recurrent or progressive ependymoma were treated in this arm. Therapy will begin with single-agent bevacizumab 10 mg/kg given intravenously (i.v) on day 1 and day 15 (+/- 24 hours) followed by MR-perfusion/diffusion imaging within 24-48 hours following the 2nd dose of bevacizumab. The first dose of irinotecan will be given i.v following this MR-perfusion scan. Subsequently, bevacizumab and irinotecan will be given every two weeks. The irinotecan dose will depend on whether the patient is on an enzyme-inducing anticonvulsant drug (EIACD). The irinotecan dose will be 250 mg/m2 (~ 80 % of dose tolerated by adults in the Duke Phase II study of bevacizumab plus irinotecan) every two weeks for those on EIACDs. If the patient is not on an EIACD, the starting dose will be 125 mg/m2.
- Low Grade Glioma: Recurrent low grade glioma(Stratum E):The only patients with recurrent low grade glioma were treated in this arm. Therapy will begin with single-agent bevacizumab 10 mg/kg given intravenously (i.v) on day 1 and day 15 (+/- 24 hours) followed by MR-perfusion/diffusion imaging within 24-48 hours following the 2nd dose of bevacizumab. The first dose of irinotecan will be given i.v following this MR-perfusion scan. Subsequently, bevacizumab and irinotecan will be given every two weeks. The irinotecan dose will depend on whether the patient is on an enzyme-inducing anticonvulsant drug (EIACD). The irinotecan dose will be 250 mg/m2 (~ 80 % of dose tolerated by adults in the Duke Phase II study of bevacizumab plus irinotecan) every two weeks for those on EIACDs. If the patient is not on an EIACD, the starting dose will be 125 mg/m2.
Arm/Group | High-grade Gliomas | Brain Stem Tumors | Ependymoma | Low Grade Glioma
Number analyzed (Participants) | 17 | 10 | 11 | 29
Ratio | -0.34 (0.085) [-0.91 to 0.26] | -0.17 [-0.60 to 0.51] | 0.11 [-0.23 to 1.38] | -0.11 [-0.89 to 0.52]

8. Secondary Outcome: Association of Log-transformed Tumor Volume Based on FLAIR With Progression-free Survival (PFS) Using Hazard Ratio Estimates
Description: Using Cox proportional hazards models, the association of tumor volume based on FLAIR images with PFS will be investigated for those strata that have a sufficient number of participants with volume FLAIR measurements. Volumetric magnetic resonance imaging is performed to investigate surrogate markers of tumor growth. Volume FLAIR measurements were longitudinal. As we are not comparing the strata, analyses will be done in each stratum separately, and thus we cannot report the Cox model results in the Statistical Analysis section. We consider these estimates 'descriptive' within each stratum. In this analysis, the hazard ratio is a relative measure of likelihood that a study participant experiences the event of interest compared to another participant who has a one-unit lower Log-transformed tumor volume based on FLAIR. The Cox survival model provides the mean hazard ratio along with its 95% confidence interval, which we report below.
Time Frame: From start of treatment until the earliest of progressive disease, death, second malignancy or off study OR up to 2 years
Population: Patients had Flair volume at Pre-treatment and at least one on treatment.
Measure: Mean (95% Confidence Interval); unit: Hazard Ratio
Arm/Group | High-grade Gliomas | Brain Stem Tumors
Number analyzed (Participants) | 13 | 12
Hazard Ratio | 1.47 [0.79 to 2.77] | 1.76 [0.65 to 4.75]

9. Secondary Outcome: Association of Log-transformed Tumor Enhancing Volume With Progression-free Survival (PFS) Using Hazard Ratio Estimates
Description: Using Cox Proportional hazards Models, the association of Log-transformed tumor enhancing volume with progression-free survival will be investigated. Volumetric magnetic resonance (MR) imaging is performed to investigate surrogate markers of tumor growth. Tumor enhancing volumes were longitudinal. As we are not comparing the strata or study arms, analyses will be done in each stratum separately, and thus we cannot report the Cox model results in the Statistical Analysis section and we consider these estimates 'descriptive' within each stratum. In this analysis, the hazard ratio is a relative measure of likelihood that a study participant experiences the event of interest compared to another participant who has a one-unit lower Log-transformed tumor enhancing volume. The Cox survival model provides the mean hazard ratio along with its 95% confidence interval, which we report below.
Time Frame: From start of treatment until the earliest of progressive disease, death, second malignancy or off study, OR up to 2 years
Population: Patients had tumor enhancing volume at Pre-treatment and at least one on treatment.
Measure: Mean (95% Confidence Interval); unit: Hazard Ratio
Groups:
- Brain Stem Tumors: Recurrent,progressive or refractory instrinsic brain stem tumors(Stratum B):The only patients with recurrent, progressive or refractory brain stem tumors were treated in this arm. Therapy will begin with single-agent bevacizumab 10 mg/kg given intravenously (i.v) on day 1 and day 15 (+/- 24 hours) followed by MR-perfusion/diffusion imaging within 24-48 hours following the 2nd dose of bevacizumab. The first dose of irinotecan will be given i.v following this MR-perfusion scan. Subsequently, bevacizumab and irinotecan will be given every two weeks. The irinotecan dose will depend on whether the patient is on an enzyme-inducing anticonvulsant drug (EIACD). The irinotecan dose will be 250 mg/m2 (~ 80 % of dose tolerated by adults in the Duke Phase II study of bevacizumab plus irinotecan) every two weeks for those on EIACDs. If the patient is not on an EIACD, the starting dose will be 125 mg/m2.
Arm/Group | High-grade Gliomas | Brain Stem Tumors
Number analyzed (Participants) | 15 | 16
Hazard Ratio | 1.65 [0.802 to 3.39] | 1.16 [0.597 to 2.27]

10. Secondary Outcome: Association of Log-transformed Volume of Cystic Necrosis With Progression-free Survival (PFS) Using Hazard Ratio Estimates
Description: Using Cox Proportional Hazards Models, the association of cystic necrosis with progression-free survival will be investigated. Volumetric magnetic resonance (MR) imaging is performed to investigate surrogate markers of tumor growth. Volumes of cystic necrosis were longitudinal. As we are not comparing the strata or study arms, analyses will be done in each stratum separately, and thus we cannot report the Cox model results in the Statistical Analysis section and we consider these estimates 'descriptive' within each stratum. In this analysis, the hazard ratio is a relative measure of likelihood that a study participant experiences the event of interest compared to another participant who has a one-unit lower Log-transformed tumor volume based on cystic necrosis. The Cox survival model provides the mean hazard ratio along with its 95% confidence interval, which we report below.
Time Frame: as for outcome 9
Population: Patients had volume of cystic necrosis at Pre-treatment and at least one on treatment.
Measure: Mean (95% Confidence Interval); unit: Hazard Ratio
Arm/Group | High-grade Gliomas | Brain Stem Tumors
Number analyzed (Participants) | 15 | 16
Hazard Ratio | 2.56 [0.89 to 7.41] | 1.09 [0.28 to 4.21]

11. Secondary Outcome: Association of Log-transformed Tumor Diffusion Ratio With Progression-free Survival (PFS) Using Hazard Ratio Estimates
Description: Using Cox Proportional Hazards Models, the association of tumor diffusion ratios with progression-free survival will be investigated. Magnetic resonance (MR) diffusion imaging is performed to investigate surrogate markers of tumor growth. Tumor diffusion ratios were longitudinal. As we are not comparing the strata or study arms, analyses will be done in each stratum separately, and thus we cannot report the Cox model results in the Statistical Analysis section. And we consider these estimates 'descriptive' within each stratum. In this analysis, the hazard ratio is a relative measure of likelihood that a study participant experiences the event of interest compared to another participant who has a one-unit lower Log-transformed tumor diffusion ratio. The Cox survival model provides the mean hazard ratio along with its 95% confidence interval, which we report below.
Time Frame: From start of treatment until the earliest of progressive disease, death, second malignancy or off study
Population: Patients had diffusion ratio at pre-treatment scans and at least one on treatment scans.
Measure: Mean (95% Confidence Interval); unit: Hazard Ratio
Arm/Group | High-grade Gliomas | Brain Stem Tumors
Number analyzed (Participants) | 17 | 14
Hazard Ratio | 4.41 [0.15 to 131] | 1.82 [0.21 to 15.9]

12. Secondary Outcome: Association of Log-transformed Tumor Perfusion Ratio With Progression-free Survival (PFS) Using Hazard Ratio Estimates
Description: Using Cox Proportional Hazards Models, the association of tumor perfusion ratio with progression-free survival will be investigated. Magnetic resonance (MR) perfusion imaging is performed to investigate surrogate markers of tumor growth. Tumor perfusion ratios were longitudinal. As we are not comparing the strata or study arms, analyses will be done in each stratum separately, and thus we cannot report the Cox model results in the Statistical Analysis section. We consider these estimates 'descriptive' within each stratum. In this analysis, the hazard ratio is a relative measure of likelihood that a study participant experiences the event of interest compared to another participant who has a one-unit lower Log-transformed tumor volume perfusion ratio. The Cox survival model provides the mean hazard ratio along with its 95% confidence interval, which we report below.
Time Frame: as for outcome 9
Population: The analyses cannot be performed with the Cox proportional hazard model since there are no sufficient measurements of perfusion ratio and events.
Arm/Group | High-grade Gliomas | Brain Stem Tumors
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Volume of Distribution
Description: Blood specimens were collected on the days listed for pharmacokinetic studies for Bevacizumab. These specimens were analyzed to produce steady-state plasma Bevacizumab concentration-time data in study participants. The concentration-time data were analyzed to provide an estimate of the volume of distribution. The data were collected but the analyses of the PK data were conducted by Genentech using a broader cohort of pediatric patients from multiple trials in the paper "Bevacizumab dosing strategy in paediatric cancer patients based on population pharmacokinetic analysis with external validation" published by British Journal of Clinical Pharmacology ,2016 volume 81(1):148-160. The estimates of the volume of distribution were calculated by the model described in the paper.
Time Frame: Baseline, Course 1 Day 1, Course 1 Day 15, Course 2 Day 1, Course 3 Day 1, Course 4 Day 1, and Course 5 Day 1
Population: The study participants across the strata (stratum A, stratum B, stratum C, stratum D, and stratum E) were combined for this secondary objective. The number of participants with available data.
Measure: Mean (Standard Deviation); unit: ml
Groups:
- Combined All Strata: High-grade Gliomas(stratum A), Medulloblastoma (stratum B), Brain Stem Tumors (stratum C), Ependymoma (stratum D), and Low Grade Glioma (stratum E) were combined for this secondary objective.
Arm/Group | Combined All Strata
Number analyzed (Participants) | 76
ml | 1729 (736.9)

14. Secondary Outcome: Systemic Clearance
Description: Blood specimens were collected on the days listed for pharmacokinetic studies for Bevacizumab. These specimens were analyzed to produce steady-state plasma Bevacizumab concentration-time data in study participants. The concentration-time data were analyzed to provide an estimate of the systemic clearance. The data were collected but the analyses of the PK data were conducted by Genentech using a broader cohort of pediatric patients from multiple trials in the paper "Bevacizumab dosing strategy in paediatric cancer patients based on population pharmacokinetic analysis with external validation" published by British Journal of Clinical Pharmacology, 2016 volume 81(1):148-160. The estimates of the systemic clearance were calculated by the model described in the paper.
Time Frame: Baseline, Course 1 Day 1, Course 1 Day 15, Course 2 Day 1, Course 3 Day 1, Course 4 Day 1, and Course 5 Day 1
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ml/h
Arm/Group | Combined All Strata
Number analyzed (Participants) | 39
ml/h | 9.43 (4.70)

15. Secondary Outcome: Terminal Half-life
Description: Blood specimens were collected on the days listed for pharmacokinetic studies for Bevacizumab. These specimens were analyzed to produce steady-state plasma Bevacizumab concentration-time data in study participants. The concentration-time data were analyzed to provide an estimate of the PK parameters. The data were collected but the analyses of the PK data were conducted by Genentech using a broader cohort of pediatric patients from multiple trials in the paper "Bevacizumab dosing strategy in paediatric cancer patients based on population pharmacokinetic analysis with external validation" published by British Journal of Clinical Pharmacology,2016 volume 81(1):148-160. The estimates of the terminal half-life were calculated by the method described in the paper.
Time Frame: Baseline, Course 1 Day 1, Course 1 Day 15, Course 2 Day 1, Course 3 Day 1, Course 4 Day 1, and Course 5 Day 1
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Combined All Strata
Number analyzed (Participants) | 39
hours | 125.2 (5.80)

16. Secondary Outcome: Change in Vascular Endothelial Growth Factor Receptor-2 (VEGF-R2) Expression in Peripheral Blood Mononuclear Cells (PBMC) From Baseline to Day-15
Description: The change in VEGF-R2 was calculated from baseline to the time of the 2nd dose (values of 24-48 hours after the 2nd dose at Day 15 - values of pre-dose 1 Day1, i.e., baseline). VEGF-R2 is measured in the relative phosphorylation score which is generated as a ratio of normalized phosphorylated VEGF-R2 versus normalized total VEGF-R2 protein.
Time Frame: Baseline and 24-48 hours after the 2nd dose of Bevacizumab in course 1
Measure: Median (Full Range); unit: Ratio
Groups:
- Brain Stem Tumors: Recurrent, progressive or refractory intrinsic brain stem tumors(Stratum B): The only patients with Recurrent, progressive or refractory brain stem tumors were treated in this arm. Therapy will begin with single-agent bevacizumab 10 mg/kg given intravenously (i.v) on day 1 and day 15 (+/- 24 hours) followed by MR-perfusion/diffusion imaging within 24-48 hours following the 2nd dose of bevacizumab. The first dose of irinotecan will be given i.v following this MR-perfusion scan. Subsequently, bevacizumab and irinotecan will be given every two weeks. The irinotecan dose will depend on whether the patient is on an enzyme-inducing anticonvulsant drug (EIACD). The irinotecan dose will be 250 mg/m2 (~ 80 % of dose tolerated by adults in the Duke Phase II study of bevacizumab plus irinotecan) every two weeks for those on EIACDs. If the patient is not on an EIACD, the starting dose will be 125 mg/m2.
- Medulloblastoma: Recurrent or progressive medulloblastoma(Stratum C):The only patients with recurrent, progressive medulloblastoma were treated in this arm. Therapy will begin with single-agent bevacizumab 10 mg/kg given intravenously (i.v) on day 1 and day 15 (+/- 24 hours) followed by MR-perfusion/diffusion imaging within 24-48 hours following the 2nd dose of bevacizumab. The first dose of irinotecan will be given i.v following this MR-perfusion scan. Subsequently, bevacizumab and irinotecan will be given every two weeks. The irinotecan dose will depend on whether the patient is on an enzyme-inducing anticonvulsant drug (EIACD). The irinotecan dose will be 250 mg/m2 (~ 80 % of dose tolerated by adults in the Duke Phase II study of bevacizumab plus irinotecan) every two weeks for those on EIACDs. If the patient is not on an EIACD, the starting dose will be 125 mg/m2.
Arm/Group | High-grade Gliomas | Brain Stem Tumors | Medulloblastoma | Ependymoma | Low Grade Glioma
Number analyzed (Participants) | 4 | 5 | 3 | 5 | 4
Ratio | -0.37 [-2.62 to 0.82] | -0.21 [-5.11 to 0.12] | -0.003 [-0.136 to 0.937] | 0.24 [-8.87 to 0.36] | 1.70 [-0.89 to 20.55]

17. Secondary Outcome: Descriptive Statistics for the Changes in Vascular Endothelial Growth Factor Receptor-2 (VEGF-R2) Expression in Peripheral Blood Mononuclear Cells (PBMC) Concurrently Measured With the Changes in Perfusion From Magnetic Resonance Imaging
Description: The changes in VEGF-R2 are calculated by values at Day 15 minus values at baseline for the patients who had the changes in perfusion from magnetic resonance perfusion imaging. The purpose of reporting descriptive statistics of changes of VEGF-R2 is to provide the information for the correlation coefficients in Section 19.
Time Frame: Baseline and Day 15 (after 2 doses of Bevacizumab) of course 1
Population: The analyses are performed for the patients who had the changes in both VEGF-R2 and perfusion.
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | High-grade Gliomas | Brain Stem Tumors
Number analyzed (Participants) | 3 | 5
Ratio | -1.12 (0.78) | -1.20 (0.99)

18. Secondary Outcome: Descriptive Statistics for the Change of Perfusion in Magnetic Resonance Imaging Concurrently Measured With the Change in Vascular Endothelial Growth Factor Receptor-2 (VEGF-R2) Expression in Peripheral Blood Mononuclear Cells (PBMC)
Description: The change of perfusion in magnetic resonance imaging is calculated by taking the difference between the Day-15 measurements and the Baseline measurements for patients who had the changes of VEGF-R2. The purpose of reporting the descriptive statistics is to provide the information for the correlation coefficients reported in the next section, Section 19. MR perfusion ratio is the ratio of the perfusion measurements in the tumor and the perfusion measurerement in comparative frontal while matter, which is the comparative healthy part of the brain.
Time Frame: Baseline and Day 15 (after 2 doses of Bevacizumab) of course 1
Population: The analyses are performed for the patients who had the changes in both VEGF-R2 and perfusion.
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | High-grade Gliomas | Brain Stem Tumors
Number analyzed (Participants) | 3 | 5
Ratio | -1.60 (1.18) | -1.54 (0.87)

19. Secondary Outcome: Correlation of the Change in Vascular Endothelial Growth Factor Receptor-2 (VEGF-R2) Expression in Peripheral Blood Mononuclear Cells (PBMC) From Baseline With the Change in Perfusion From Magnetic Resonance Imaging
Description: Spearman correlation coefficient is used to measure the correlation of the changes in VEGF-R2 with the changes in perfusion ratios. The changes are calculated by values at Day 15 minus values at baseline for VEGF-2 in Section 17 above and perfusion in Section 18 above, respectively. The correlation coefficients are reported in each stratum separately.
Time Frame: Baseline and Day 15 (after 2 doses of Bevacizumab) of course 1
Population: The analyses are performed for the patients who had the changes in both VEGF-R2 and perfusion.
Measure: Number; unit: Correlation Coefficient
Arm/Group | High-grade Gliomas | Brain Stem Tumors
Number analyzed (Participants) | 3 | 5
Correlation Coefficient | 0.5 (0.61) | -0.50 (0.27)

20. Secondary Outcome: Number of Patients With High Hypoxia Inducible Factor-2alpha Expression at Baseline
Description: The expression of Hypoxia inducible factor-2α, carbonic anhydrase IX (CA9), VEGF-A, and VEGF-R2 will be estimated by immunohistochemistry of paraffin sections in the medulloblastoma,ependymoma and low grade glioma strata. Reported separately for each stratum.
Time Frame: Baseline
Population: Only strata were reported, in which the patients had tissue samples available.
Measure: Number; unit: participants
Arm/Group | Medulloblastoma | Ependymoma | Low Grade Glioma
Number analyzed (Participants) | 4 | 5 | 17
participants | 0 | 3 | 7

21. Secondary Outcome: Number of Patients With High Carbonic Anhydrase 9 Expression at Baseline
Description: as for outcome 20
Time Frame: Baseline
Population: Only strata were reported, in which the patients had tissue samples available.
Measure: Number; unit: participants
Arm/Group | Medulloblastoma | Ependymoma | Low Grade Glioma
Number analyzed (Participants) | 4 | 5 | 17
participants | 0 | 4 | 2

22. Secondary Outcome: Number of Patients With High VEGF-A Expression at Baseline
Description: as for outcome 20
Time Frame: Baseline
Population: Only strata were reported, in which the patients had tissue samples available.
Measure: Number; unit: participants
Arm/Group | Medulloblastoma | Ependymoma | Low Grade Glioma
Number analyzed (Participants) | 4 | 5 | 18
participants | 2 | 5 | 16

23. Secondary Outcome: Number of Patients With High VEGF-R2 Expression at Baseline
Description: as for outcome 20
Time Frame: Baseline
Population: Only strata were reported, in which the patients had tissue samples available.
Measure: Number; unit: participants
Arm/Group | Medulloblastoma | Ependymoma | Low Grade Glioma
Number analyzed (Participants) | 4 | 5 | 18
participants | 4 | 4 | 13

24. Secondary Outcome: Progression-free Survival Hazard Ratio by Hypoxia Inducible Factor-2alpha Expression
Description: The association of hypoxia inducible factor-2alpha expression with progression-free survival will be investigated for those strata that have a sufficient number of participants with hypoxia inducible factor-2alpha measurements. The hazard ratio was reported for patients who had hypoxia inducible factor-2alpha expression.
Time Frame: From start of treatment until the earliest of progressive disease, death, second malignancy or off study
Population: The number of patients in strata C and D was not sufficient to perform the analysis exploring the association of hypoxia inducible factor-2alpha expression with progression-free survival. Thus the association analysis was performed for the patients in Stratum E only.
Measure: Number (95% Confidence Interval); unit: Hazard Ratio
Arm/Group | Low Grade Glioma
Number analyzed (Participants) | 17
Hazard Ratio | 1.36 [0.364 to 5.083]

25. Secondary Outcome: Progression-free Survival Hazard Ratio by Carbonic Anhydrase 9 (CA9) Expression
Description: The association of CA9 expression with progression-free survival will be investigated for those strata that have a sufficient number of participants with CA9 measurements.
Time Frame: From start of treatment until the earliest of progressive disease, death, second malignancy or off study
Population: Only the number of patients in strata E was sufficient to perform the analysis exploring the association of carbonic anhydrase 9 (CA9) expression with progression-free survival.
Measure: Number (95% Confidence Interval); unit: Hazard Ratio
Arm/Group | Low Grade Glioma
Number analyzed (Participants) | 17
Hazard Ratio | 0.705 [0.089 to 5.598]

26. Secondary Outcome: Progression-free Survival Hazard Ratio by VEGF-A Expression
Description: The association of VEGF-A expression with progression-free survival will be investigated for those strata that have a sufficient number of participants with VEGF-A measurements.
Time Frame: From start of treatment until the earliest of progressive disease, death, second malignancy or off study
Population: Only the number of patients in strata E was sufficient to perform the analysis exploring the association of VEGF-A expression with progression-free survival.
Measure: Number (95% Confidence Interval); unit: Hazard Ratio
Arm/Group | Low Grade Glioma
Number analyzed (Participants) | 18
Hazard Ratio | 0.091 [0.006 to 1.510]

27. Secondary Outcome: Progression-free Survival Hazard Ratio by VEGF-R2 Expression
Description: The association of VEGF-R2 expression with progression-free survival will be investigated for those strata that have a sufficient number of participants with VEGF-R2 measurements.
Time Frame: From start of treatment until the earliest of progressive disease, death, second malignancy or off study
Population: Only the number of patients in strata E was sufficient to perform the analysis exploring the association of VEGF-R2 expression with progression-free survival.
Measure: Number (95% Confidence Interval); unit: Hazard Ratio
Arm/Group | Low Grade Glioma
Number analyzed (Participants) | 18
Hazard Ratio | 0.632 [0.161 to 2.482]

ADVERSE EVENTS:
Time Frame: 2 Years
Groups:
- PBTC-022: Children with recurrent,progressive,or refractory malignant gliomas, diffuse/intrinsic brain stem gliomas, medulloblastomas and low grade gliomas
Arm/Group | PBTC-022
Serious Adverse Events (participants affected / at risk) | 37/92
Other Adverse Events (participants affected / at risk) | 91/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PBTC-022 (N=92)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (3)
Alkalosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dysphasia (Nervous system disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Leukoencephalopathy (Nervous system disorders) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (2)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 2 (2)
Neutrophil count decreased (Investigations) | 3 (3)
Personality change (Psychiatric disorders) | 1 (1)
Platelet count decreased (Investigations) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Psychosis (Psychiatric disorders) | 1 (1)
Seizure (Nervous system disorders) | 5 (8)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3)
Weight loss (Investigations) | 2 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PBTC-022 (N=92)
Acidosis (Metabolism and nutrition disorders) | 11 (22)
Alanine aminotransferase increased (Investigations) | 28 (37)
Alkaline phosphatase increased (Investigations) | 6 (13)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 13 (16)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (8)
Anorexia (Metabolism and nutrition disorders) | 19 (25)
Aspartate aminotransferase increased (Investigations) | 32 (50)
Ataxia (Nervous system disorders) | 11 (16)
Blood bilirubin increased (Investigations) | 7 (13)
Constipation (Gastrointestinal disorders) | 16 (21)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (15)
Creatinine increased (Investigations) | 6 (11)
Diarrhea (Gastrointestinal disorders) | 45 (113)
Dizziness (Nervous system disorders) | 10 (13)
Extraocular muscle paresis (Eye disorders) | 5 (5)
Fever (General disorders) | 16 (23)
GGT increased (Investigations) | 6 (8)
Hyperglycemia (Metabolism and nutrition disorders) | 17 (24)
Hyperkalemia (Metabolism and nutrition disorders) | 9 (10)
Hypermagnesemia (Metabolism and nutrition disorders) | 17 (30)
Hypernatremia (Metabolism and nutrition disorders) | 7 (8)
Hypertension (Vascular disorders) | 37 (74)
Hypoalbuminemia (Metabolism and nutrition disorders) | 15 (22)
Hypocalcemia (Metabolism and nutrition disorders) | 19 (38)
Hypoglycemia (Metabolism and nutrition disorders) | 10 (14)
Hypokalemia (Metabolism and nutrition disorders) | 24 (32)
Hypomagnesemia (Metabolism and nutrition disorders) | 11 (22)
Hyponatremia (Metabolism and nutrition disorders) | 11 (20)
Hypophosphatemia (Metabolism and nutrition disorders) | 21 (41)
Intracranial hemorrhage (Nervous system disorders) | 10 (10)
Lymphocyte count decreased (Investigations) | 42 (92)
Nausea (Gastrointestinal disorders) | 52 (129)
Neutrophil count decreased (Investigations) | 27 (57)
Platelet count decreased (Investigations) | 11 (25)
Proteinuria (Renal and urinary disorders) | 20 (61)
Rash acneiform (Skin and subcutaneous tissue disorders) | 6 (8)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 16 (21)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 5 (5)
Tremor (Nervous system disorders) | 6 (6)
Urinary retention (Renal and urinary disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 56 (282)
White blood cell decreased (Investigations) | 44 (85)

LIMITATIONS AND CAVEATS:
Neuroimaging data capturing Volume Enhancing and Perfusion Ratio was so limited to run any statistical model. Similarly, due to limited data, some PK and Biology objectives were not able to be addressed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less